CLINICAL TRIAL: NCT04669236
Title: Promoting Healthy Sleep in Adolescents: a Participatory Health Research Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B670201630466
Record Dates: First submitted 2018-11-12; First posted 2020-12-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Sleep
Keywords: Sleep behaviour; Adolescents; Participatory health research; Intervention

STUDY DESIGN:
Intervention Model Description: Pre, post and follow-up testing with 3 intervention and 6 control schools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention promoting healthy sleep behaviour in adolescents based on a participatory health research approach. Based on participatory session, the pupils of the action group will develop the intervention. They will participate in every step of the development to maximize their input.
  Interventions: Behavioral: Intervention to promote healthy sleep behavior
- Control group (No Intervention): Participants in the control group will receive no intervention.

INTERVENTIONS:
Behavioral: Intervention to promote healthy sleep behavior — An action group (6 - 8 pupils) was conducted at each school. Brainstorm sessions about effective strategies to change sleeping behavior in this population were held. Strategies, perceived as effective by the target population, will be summarized in an overview. Also feedback of adolescent, who are not part of the action group, will be asked. After feedback, the intervention will be developed by the intervention schools. Thereby, three different intervention strategies will be implemented and tested (one intervention at each school) to meet the individuals needs of each school. The action groups will develop the intervention materials during sessions this year. Afterwards, they will implement the intervention themselves in collaboration with teachers of the school and the researchers.
  Arms: Intervention group

SUMMARY:
Adolescent sleep deprivation is becoming increasingly recognized internationally as a significant health concern. This project will be the first to use a unique approach of actively involving adolescents as real life experts in the development of interventions to improve sleep behaviour (using a participatory health research methodology) and to evaluate the effectiveness of these interventions (using a randomised controlled trial).

DETAILED DESCRIPTION:
The project will develop an intervention to promote healthy sleep behaviour in adolescents. The intervention will be based on a participatory health research approach to promote healthy sleep behaviour in adolescents. Because healthy sleep behaviour is associated with a healthy lifestyle overall, the intervention will additionally focus on healthy eating patterns, sedentary behaviour and physical activity. In order to become the most effective intervention, adolescents will participate during every step of the intervention development.

Three school in Flanders are contributing to this project on a voluntary basis. All adolescents age 13 to 15 of the intervention schools were invited to participate in the study by an informative session at the school, where they were informed about the importance of their involvement in the study and the aim of the intervention. The adolescents who gave their consent, were invited to participate in a workshop were skills needed for participatory research were trained. Afterwards, an action group (6 - 8 pupils) was conducted at each school. Brainstorm sessions about effective strategies to change sleeping behavior in this population. Strategies, perceived as effective by the target population, will be summarized in an overview. Also feedback of adolescent, who are not part of the action group, will be asked. After feedback, the intervention will be developed by the intervention schools. Thereby, three different intervention strategies will be implemented and tested (one intervention at each school) to meet the individuals needs of each school. Right now, the action groups are busy conducting the intervention materials during a weekly 1-hour session. This session is accompanied by two researchers to provoke brainstorm sessions and creativity. The researchers facilitate the process, stimulates creativity, organize and keep track of the feasibility of ideas. After the development of intervention materials, the intervention will be implemented in the school by the adolescents themselves, in collaboration with teachers and the two researchers.

Overall, can be stated that a group oriented approach will be used during the whole intervention. For example, plenary speakers will give information about sleep hygiene, physical activity breaks will be introduced, sleep behaviour will be discussed in class, active transport will be stimulated, a campaign on social media will be started, and informative flyers/posters about sleep, screen time, physical activity and nutrition will be spread in the close neighborhood, a competition between class groups will be started (based on objective data collected using activity trackers).

The intervention will be analysed using a clustered randomized controlled trial, including three intervention schools and six control schools. These schools were recruited in Flanders, the Northern part of Belgium, via convenience sampling. The head of each school was contacted via telephone. When the head of the school gave consent, all adolescents age 13 - 15 and their parents were invited to participate in this study. All adolescents who gave their consent, were pre-tested (between November 2017 and January 2018). The pre-test included a questionnaire investigating determinants of sleep and a wearable activity tracker to objectively measure the sleep duration. The questionnaires were developed based on the 'Munich ChronoType Questionnaire', 'The School Sleep Habits Survey', 'Sleep Knowledge Questionnaire', 'Sleep Hygiene Index' and 'Paediatric Daytime Sleepiness Scale'. Focus groups were organized to determine relevant determinants. The understandability of the questionnaire was tested with the 'Thinking aloud protocol' and validation testing was performed. After implementing the intervention at the intervention schools, an effect-evaluation will be conducted based on a pre-,post and follow-up testing and a process evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 and 16 years old
* Dutch speaking
* Education: ASO (General Secondary Education), TSO (Technical Secondary Education) or BSO (Vocational Secondary Education)

Exclusion Criteria:

* Having a sleeping disorder
* BUSO (Special Secondary Education)

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2044 (Actual)
Dates: Start 2017-06-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Sleep duration as assesed by the Munich Chronotype Questionnaire for children | 2 years
  to ask about students' sleep habits over the past 2 weeks, differentiating between sleep on school nights (Sunday to Thursday) and weekend nights (Friday and Saturday). Students will be asked to report their typical go to bed time, lights-out time, sleep onset latency, total sleep time, wake-up time, and out of bed time. This questionnaire showed good validity against objective sleep measures (i.e., actigraphy).
Sleep quality as assesed by the short Adolescent Sleep Wake Scale | 2 years
  10 questions on sleep quality and sleep habbits, topics are: going to bed, during the night and waking up

SECONDARY OUTCOMES:
Sleep knowledge | 2 years
  Sleep knowledge will be measured using a Sleep Knowledge Questionnaire consisting of 15 questions with a true/false response format. This questionnaire has shown to be sensitive to changes and to offer a degree of discriminant validity; however, the test-retest reliability is unknown and will be tested at the start of this project.
Sleep hygiene | 2 years
  Sleep hygiene will be assessed using the Sleep Hygiene Index including 13 items scored on 5-point Likert-type scale with answers (1) ranging from always to never (5). A sum score can be made of all questions to obtain a total score. The higher the total score, the better the sleep hygiene. The internal consistency of this scale is found to be acceptable and test-retest reliability is good.
Daytime sleepiness | 2 years
  Daytime sleepiness will be measured by the validated Paediatric Daytime Sleepiness Scale. This scale contains eight items about aspects of daytime sleepiness experienced by students (e.g., How often do you get sleepy or drowsy while doing your homework?). Answers range from never (0) to always (4) on 5-point Likert-type scale. For total score, a sum score should be made of all answers. Abnormal values: 6th and 7th grade >26, 8th grade >30.
Socio-demographic and theory-based psychosocial correlates | 2 years
  Socio-demographic and theory-based psychosocial correlates of sleep behaviour will be measured by a self-developed questionnaire based on existing questionnaires assessing correlates of health behaviour used in previous studies of our research group. The questionnaire will be pilot-tested on comprehension and psychometrics at the start of this project.

CONTACTS AND LOCATIONS:
Overall Officials: Benedicte Deforche, Study Director — University Ghent
Locations (1):
- Ghent University-Public Health Department, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vandendriessche A, Deforche B, Dhondt K, Verloigne M, Van Cauwenberg J. Effect evaluation of a participatory developed school-based healthy sleep intervention for adolescents. Health Psychol. 2025 Apr;44(4):380-390. doi: 10.1037/hea0001443. Epub 2025 Jan 27. PMID 39869691